CLINICAL TRIAL: NCT06799065
Title: A Phase 1/2, Open-Label, Dose-Escalation and Expansion First-In-Human Study of ATX-295, an Oral Inhibitor of the Kinesin Motor Protein KIF18A, in Patients With Locally Advanced or Metastatic Solid Tumors, Including High-Grade Serous Ovarian Cancer
Brief Title: First-in-Human Study of ATX-295, an Oral Inhibitor of KIF18A, in Patients With Advanced or Metastatic Solid Tumors, Including Ovarian Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Accent Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ATX-295-001
Record Dates: First submitted 2025-01-18; First posted 2025-01-29 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Advanced Solid Tumors; Breast Cancer Recurrent; Ovarian Cancer; High-grade Serous Ovarian Carcinoma; Triple Negative Breast Cancer
Keywords: KIF; KIF18A; HGSOC; Platinum-resistant; Platinum-intolerant; Platinum-refractory
MeSH Terms: conditions — Ovarian Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dose Escalation (Experimental): Subjects will be enrolled at various doses and/or schedules of ATX-295 to identify the expansion dose(s) and RP2D
  Interventions: Drug: ATX-295
- Dose Expansion: Platinum-Resistant, -Refractory, or -Intolerant HGSOC (Experimental)
  Interventions: Drug: ATX-295

INTERVENTIONS:
Drug: ATX-295 — ATX-295 Tablets will be taken orally

SUMMARY:
The goal of this study is to identify a safe and tolerated dose of the orally administered KIF18A inhibitor ATX-295. In addition, this study will evaluate the pharmacokinetics, pharmacodynamics and preliminary antitumor activity of ATX-295 in patients with advanced solid tumors and ovarian cancer.

DETAILED DESCRIPTION:
ATX-295 is an oral drug that inhibits a protein called KIF18A, an adenosine triphosphate (ATP)-dependent, plus end-directed mitotic kinesin. KIF18A facilitates chromosomal alignment and spindle microtubule dynamics during mitosis in certain advanced solid tumors. ATX-295 has been shown preclinically to induce robust anti-tumor activity of a variety of different solid tumors, including high-grade serious ovarian cancer and triple negative breast cancer.

This is a first-in-human, Phase 1, open-label, single-arm, dose-escalation and Simon 2-Stage expansion study to evaluate the safety profile of ATX-295 and determine the recommended phase 2 dose (RP2D). In addition, the study aims to characterize the PK, PD, and preliminary anti-tumor activity of orally administered ATX-295. Exploratory objectives include examination of biomarker responses in relationship to ATX-295 exposure.

Patients with locally advanced or metastatic solid tumors will be enrolled to preliminarily assess the anti-tumor effect, and further examine the safety and PK of ATX-295 at the RP2D.

ELIGIBILITY:
Key Inclusion Criteria:

* Patients with histologically confirmed solid tumors who have locally recurrent or metastatic disease, including HGSOC
* Refractory to or relapsed after all standard therapies with proven clinical benefit, unless as deemed by the Investigator, the subject is not a candidate for standard treatment, there is no standard treatment, or the subject refuses standard treatment after expressing an understanding of all available therapies with proven clinical benefit
* For the expansion cohorts, participants must have histological confirmation of HGSOC and be determined to be platinum-resistant, platinum-refractory, or platinum-intolerant
* There is no limit to the number of prior treatment regimens
* Have measurable or evaluable disease
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1

Key Exclusion Criteria:

* Clinically unstable central nervous system (CNS) tumors or brain metastasis
* Any other concurrent anti-cancer treatment, except for hormonal blockade
* Has undergone a major surgery within 3 weeks of starting study treatment
* Medical issue that limits oral ingestion or impairment of gastrointestinal function that is expected to significantly reduce the absorption of ATX-295, however participants with a functioning distal ileostomy or colostomy may be permitted on trial
* Clinically significant (ie, active) or uncontrolled cardiovascular disease
* Need to use proton pump inhibitors on study or H2-receptor antagonists for the dose escalation portion of the study.
* Unable to transition off strong or moderate CYP3A4 inhibitors or strong inducers
* Pregnancy or intent to breastfeed or conceive a child within the projected duration of treatment

Other inclusion and exclusion criteria as defined in the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-08-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) and/or maximum tolerated dose (MTD) of ATX-295 | 12 months
  Identification of a tolerable and safe dose for expansion cohorts based on dose limiting toxicities
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) | 12 months
  Adverse events graded according to CTCAE v5.0

SECONDARY OUTCOMES:
Preliminary evidence of antitumor activity | 12 months
  Objective response rate based on RECIST v1.1
Measurement of phospho-histone H3 in pre- and post-treatment biopsies for a subset of participants (pharmacodynamic biomarker) | 12 months
Maximum observed plasma concentration of ATX-295 (Cmax) | 12 months
Calculated time to reach maximum observed plasma concentration (Tmax) | 12 months
Calculated area under the plasma concentration-time curve of ATX-295 (AUC0-t) | 12 months

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Sarasota, Florida
  - SCRI Oncology Partners, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - NEXT Virginia, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No